CLINICAL TRIAL: NCT01446237
Title: An Open-Label, 12-Week Study to Evaluate the Efficacy and Safety of the Acne System (Benzoyl Peroxide 2.5%, Salicylic Acid 0.5%) in Subjects With Acne
Brief Title: U0289-405: An Open-Label, 12-Week Study to Evaluate the Efficacy and Safety of the Acne System (Benzoyl Peroxide 2.5%, Salicylic Acid 0.5%) in Subjects With Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115576
Record Dates: First submitted 2011-07-28; First posted 2011-10-05 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acne system - benzoyl peroxide 2.5%, Salicylic Acid 0.5% (Experimental): open label - no comparator; only Acne system - benzoyl peroxide 2.5%, Salicylic Acid 0.5%
  Interventions: Other: acne system - benzoyl peroxide 2.5%, Salicyclic Acid 0.5%

INTERVENTIONS:
Other: acne system - benzoyl peroxide 2.5%, Salicyclic Acid 0.5% — over the counter acne system

SUMMARY:
This study is being conducted to obtain safety, efficacy, and satisfaction data on the combination of topical Benzoyl Peroxide (BPO) 2.5% and the topical keratolytic agent Salicylic Acid (SA) 0.5% in the treatment of moderate to severe acne. Subjects with moderate or severe acne will be asked to apply the commercially available, over-the-counter products Foam Deep Cleanser (2.5% BPO), Foam Advanced Acne Treatment (2.5% BPO), and Foam Rejuvenating Toner (0.5% SA) daily for 12 weeks. No control group or reference treatment will be included.

DETAILED DESCRIPTION:
This open-label, multicenter, study is being conducted to obtain safety, efficacy, and satisfaction data on an Acne System (Benzoyl Peroxide 2.5%, Salicylic Acid 0.5%), which includes Foam Deep Cleanser (2.5% Benzoyl Peroxide) and Foam Advanced Acne Treatment (2.5% Benzoyl Peroxide) and Foam Rejuvenating Toner (0.5% Salicylic Acid), in the treatment of moderate to severe acne. Approximately 120 male or female subjects ages 12-35 years, inclusive, with moderate or severe acne as assessed by Investigator's Global Assessment (ISGA) and lesion counts are expected to be enrolled. Subjects will be instructed to use all 3 study products as part of a complete acne treatment system; no reference therapy or control group will be included. Subjects will be instructed to apply Foam Deep Cleanser (2.5% Benzoyl Peroxide) and Foam Advnced Acne Treatment (2.5% Benzoyl Peroxide) to the face each morning and Foam Deep Cleanser (2.5% Benzoyl Peroxide) and Foam Rejuvenating Toner (0.5% Salicylic Acid) each evening over an application period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol-specific procedures are performed.
* Male or female ages 12 to 35 years, inclusive at time of consent.
* ISGA score of 3 or 4 at Baseline.
* Lesion counts meeting all of the following criteria: A: A minimum of 25 but not more than 50 facial inflammatory lesions (papules and pustules), excluding nasal lesions. B: A minimum of 20 but not more than 100 facial non-inflammatory lesions (open and closed comedones), excluding nasal lesions. C: No more than 3 facial nodular lesions (<5mm), with no cystic lesions.
* Ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study.
* Negative urine pregnancy test for females of childbearing potential.
* Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product.

Exclusion Criteria:

* Female who is pregnant, trying to become pregnant, or breast feeding.
* History of lupus, dermatomyositis, rosacea, seborrheic dermatitis, beard folliculitis, polycystic ovary syndrome, hirsutism, or perioral dermatitis. (Subjects with Seborrheic dermatitis may be enrolled if the condition has been inactive for at least 1 year and/or it does not affect the face.)
* Use of topical antibiotics on the face within the past 2 weeks or of systemic antibiotics for acne treatment within the past 4 weeks.
* Concurrent use of medications known to be photosensitizers (eg, thiazides, tetracyclines, fluoroquinolones, phenothiazines, and sulfonamides) because of the possibility of augmented photosensitivity.
* Use of topical corticosteroids on the face within the past 2 weeks or systemic corticosteroids within the past 4 weeks. Use of inhaled, intra-articular, or intra-lesional steroids other than for facial acne is acceptable.
* Use of systemic retinoids (eg, isotretinoin) within the past 6 months.
* Treatment with estrogens, including oral, implanted, injected, and topical contraceptives, androgens, or anti-androgenic agents for 12 weeks or fewer immediately prior to study enrollment. Subjects that have been treated with estrogens, as described above, androgens, or anti-androgenic agents for more than 12 consecutive weeks prior to study enrollment are allowed to enroll as long as they do not expect to change the dose or drug, or to discontinue use during the study and it has not been indicated for the treatment of acne vulgaris.
* Male with facial hair that could interfere with study assessments.
* Use of topical anti-acne medications (eg, BPO, retinoids, azelaic acid, resorcinol, sulfur and derivatives, SA, alpha or beta hydroxy acids, antioxidants, anti-wrinkle, antimicrobials, glycolic acid, abradants) within the past 2 weeks. Use of superficial facial procedures, and natural/herbal products within the past 4 weeks.
* Concomitant use of medications that are reported to exacerbate acne as these may impact efficacy assessments.
* Facial procedure (eg, blue light, chemical or laser peel, microdermabrasion) performed by aesthetician, beautician, physician, nurse, or other practitioner within the past 8 weeks.
* facial skin cancer diagnosis in preceding 12 months.
* Require or desire excessive or prolonged exposure to ultraviolet light (eg, sunlight or tanning beds) during the study.
* Dermatological disorder that in the opinion of the investigator may interfere with the accurate evaluation of the subject's facial appearance.
* Any major illness within 4 weeks before study enrollment.
* Previous use of the study products.
* Use of any investigational drug or procedure within the past 4 weeks or currently participating in another clinical study.
* Known hypersensitivity or previous allergic reaction to any of the active components of the study product.
* Any other condition which, in the judgement of the investigator, would put the subject at unacceptable risk for participation in the study.
* Current drug or alcohol abuse. (Drug screening is not required.)
* Considered unable or unlikely to attend the necessary visits.
* Employee of the investigator, clinical research organization, Stiefel, a GSK company, or GlaxoSmithKline (GSK) who is involved in the study, or an immediate family member (eg, partner, offspring, parents, siblings or sibling's offspring) of an employee who is involved in the study.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2011-06-01; Primary Completion 2011-12-01 (Actual); Study Completion 2011-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (9):
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Belleville, New Jersey
  - GSK Investigational Site, Montclair, New Jersey
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115576 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115576 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115576 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115576 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115576 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115576 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115576 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 125 participants of 12 to 35 years from 9 centers in the United States were enrolled in this 12 Week study to evaluate the efficacy and safety of the MaxClarity System in participants with acne. The study started on 23 June 2011 and completed on 14 December 2011.
Groups:
- MaxClarity: Participants were instructed to apply MaxClarity Foam Deep Cleanser (2.5 percent (Benzoyl Peroxide[BPO]) and MaxClarity Foam Advanced Acne Treatment (2.5 percent BPO) to the face each morning and MaxClarity Foam Deep Cleanser (2.5 percent BPO) and MaxClarity Foam Rejuvenating Toner (0.5 percent salicylic acid [SA]) each evening over an application period of 12 weeks.
Period: Overall Study
Arm/Group | MaxClarity
Started | 125
Completed | 115
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Groups:
- MaxClarity: Participants were instructed to apply MaxClarity Foam Deep Cleanser (2.5 percent (BPO) and MaxClarity Foam Advanced Acne Treatment (2.5 percent BPO) to the face each morning and MaxClarity Foam Deep Cleanser (2.5 percent BPO) and MaxClarity Foam Rejuvenating Toner (0.5 SA) each evening over an application period of 12 weeks.
Arm/Group | MaxClarity
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.0 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 57
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 7
  Asian | 9
  Black | 21
  Native Hawaiian or Other Pacific Islander | 1
  White | 84
  American Indian or Alaska Native/Asian | 1
  American Indian or Alaska Native/Black | 1
  Biracial | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Changes in Inflammatory (IL), Non-inflammatory (NIL), and Total Lesion (TL) Counts From Baseline to Each Study Visit
Description: The investigator assessed efficacy at Baseline (Day 1), Week 1, 2, 4, 8 and 12 by lesion counts- IL (papules and pustules), NIL (open and closed comedones), and TL. The area considered for efficacy assessments was confined to the face. The area of the face to be examined extended from the hairline to the mandible; includes the forehead, cheeks, and chin; and excludes the mouth, nasal region, periocular area, and superior and inferior eyelids. Baseline was defined at Day 1. Change from Baseline is value at indicated time point minus the Baseline value. Mean percent change from baseline at each study visit was presented.
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8, 12
Population: Intent-to-treat (ITT) population consisted of all participants that were enrolled in the study. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change in lesions
Arm/Group | MaxClarity
Number analyzed (Participants) | 125
Percent change in lesions
  IL Week 1: number analyzed (Participants) | 120
  IL Week 1 | -30.4 (25.8)
  IL Week 2: number analyzed (Participants) | 121
  IL Week 2 | -44.8 (26.4)
  IL Week 4: number analyzed (Participants) | 120
  IL Week 4 | -52.9 (27.0)
  IL Week 8: number analyzed (Participants) | 116
  IL Week 8 | -59.8 (23.7)
  IL Week 12: number analyzed (Participants) | 122
  IL Week 12 | -67.1 (22.7)
  NIL Week 1: number analyzed (Participants) | 120
  NIL Week 1 | -14.8 (24.4)
  NIL Week 2: number analyzed (Participants) | 121
  NIL Week 2 | -28.5 (24.4)
  NIL Week 4: number analyzed (Participants) | 120
  NIL Week 4 | -37.1 (30.1)
  NIL Week 8: number analyzed (Participants) | 116
  NIL Week 8 | -43.8 (29.3)
  NIL Week 12: number analyzed (Participants) | 122
  NIL Week 12 | -57.3 (25.8)
  TL Week 1: number analyzed (Participants) | 120
  TL Week 1 | -22.2 (20.6)
  TL Week 2: number analyzed (Participants) | 121
  TL Week 2 | -36.0 (21.5)
  TL Week 4: number analyzed (Participants) | 120
  TL Week 4 | -44.4 (23.6)
  TL Week 8: number analyzed (Participants) | 116
  TL Week 8 | -51.0 (23.2)
  TL Week 12: number analyzed (Participants) | 122
  TL Week 12 | -61.6 (22.0)

2. Primary Outcome: Number of Participants With a Minimum 2-grade Improvement of Investigator's Static Global Assessment (ISGA) From Baseline to Each Study Visit
Description: The investigator assessed efficacy at Baseline (Day 1), Week 1, 2, 4, 8 and 12 by ISGA scale: 0- Clear (clear skin with IL or NIL), 1- Almost clear (Rare NIL with no more than rare papules), 2- Mild (greater than Grade 1, some NIL with no more than a few IL (papules/pustules only, no nodular lesions), 3- Moderate (greater than Grade 2, up to many NIL and may have some IL, but no more than one small nodular lesion), 4- Severe (greater than Grade 3, up to many NIL and IL, but no more than a few nodular lesions) and 5- Very severe (Many NIL and IL and more than a few nodular lesions. May have cystic lesions). Baseline was defined at Day 1. Change from Baseline is value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8, 12
Population: ITT population. Only those participants with data available at that particular time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | MaxClarity
Number analyzed (Participants) | 125
Participants
  Week 1: number analyzed (Participants) | 120
  Week 1 | 3
  Week 2: number analyzed (Participants) | 121
  Week 2 | 6
  Week 4: number analyzed (Participants) | 120
  Week 4 | 12
  Week 8: number analyzed (Participants) | 116
  Week 8 | 19
  Week 12: number analyzed (Participants) | 122
  Week 12 | 31

3. Primary Outcome: Number of Participants With ISGA Score of 0 (Clear) or 1 (Almost Clear) at Each Study Visit
Description: The investigator assessed efficacy at baseline (Day 1), Week 1, 2, 4, 8 and 12 by ISGA scale: 0- Clear (clear skin with IL or NIL), 1- Almost clear (Rare NIL with no more than rare papules), 2- Mild (greater than Grade 1, some NIL with no more than a few IL (papules/pustules only, no nodular lesions), 3- Moderate (greater than Grade 2, up to many NIL and may have some IL, but no more than one small nodular lesion), 4- Severe (greater than Grade 3, up to many NIL and IL, but no more than a few nodular lesions) and 5- Very severe (Many NIL and IL and more than a few nodular lesions. May have cystic lesions).
Time Frame: Week 1, 2, 4, 8 and 12
Population: ITT population.
Measure: Number; unit: Participants
Arm/Group | MaxClarity
Number analyzed (Participants) | 125
Participants
  Week 1 | 1
  Week 2 | 2
  Week 4 | 4
  Week 8 | 10
  Week 12 | 20

4. Secondary Outcome: Absolute Change in IL, NIL, and TL Count From Baseline to Each Study Visit
Description: The investigator assessed efficacy at Baseline (Day 1), Week 1, 2, 4, 8 and 12 by lesion counts- IL (papules and pustules), NIL (open and closed comedones), and TL. The area considered for efficacy assessments was confined to the face. The area of the face to be examined extends from the hairline to the mandible; includes the forehead, cheeks, and chin; and excludes the mouth, nasal region, periocular area, and superior and inferior eyelids. Baseline was defined at Day 1. Change from Baseline is value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8, 12
Population: ITT population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | MaxClarity
Number analyzed (Participants) | 125
Lesions
  IL Week 1: number analyzed (Participants) | 120
  IL Week 1 | -9.6 (8.2)
  IL Week 2: number analyzed (Participants) | 121
  IL Week 2 | -14.3 (8.9)
  IL Week 4: number analyzed (Participants) | 120
  IL Week 4 | -16.9 (9.3)
  IL Week 8: number analyzed (Participants) | 116
  IL Week 8 | -18.9 (8.0)
  IL Week 12: number analyzed (Participants) | 122
  IL Week 12 | -21.4 (8.2)
  NIL Week 1: number analyzed (Participants) | 120
  NIL Week 1 | -7.4 (12.1)
  NIL Week 2: number analyzed (Participants) | 121
  NIL Week 2 | -13.4 (13.5)
  NIL Week 4: number analyzed (Participants) | 120
  NIL Week 4 | -17.6 (15.4)
  NIL Week 8: number analyzed (Participants) | 116
  NIL Week 8 | -20.1 (16.3)
  NIL Week 12: number analyzed (Participants) | 122
  NIL Week 12 | -25.6 (15.3)
  TL Week 1: number analyzed (Participants) | 120
  TL Week 1 | -17.0 (16.6)
  TL Week 2: number analyzed (Participants) | 121
  TL Week 2 | -27.7 (18.8)
  TL Week 4: number analyzed (Participants) | 120
  TL Week 4 | -34.5 (20.3)
  TL Week 8: number analyzed (Participants) | 116
  TL Week 8 | -38.9 (20.4)
  TL Week 12: number analyzed (Participants) | 122
  TL Week 12 | -47.0 (19.8)

5. Secondary Outcome: Mean Change in ISGA From Baseline to Each Study Visit
Description: as for outcome 2
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8, 12
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MaxClarity
Number analyzed (Participants) | 125
Scores on a scale
  Week 1: number analyzed (Participants) | 120
  Week 1 | -0.29 (0.51)
  Week 2: number analyzed (Participants) | 121
  Week 2 | -0.45 (0.61)
  Week 4: number analyzed (Participants) | 120
  Week 4 | -0.63 (0.69)
  Week 8: number analyzed (Participants) | 116
  Week 8 | -0.79 (0.75)
  Week 12: number analyzed (Participants) | 122
  Week 12 | -1.05 (0.78)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from screening visit, Baseline (Day 1) and up to Week 12/early termination.
Description: ITT population was used for all analyses which comprised of all participants enrolled in the study.
Arm/Group | MaxClarity
All-Cause Mortality (participants affected / at risk) | 0/125
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 12/125
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MaxClarity (N=125)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
SEASONAL ALLERGY (Immune system disorders) | 1
NASOPHARYNGITIS (Infections and infestations) | 3
ORAL HERPES (Infections and infestations) | 2
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1
POST PROCEDURAL INFECTION (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1
CONTUSION (Injury, poisoning and procedural complications) | 1
BURNING SENSATION (Nervous system disorders) | 1
OVARIAN CYST (Reproductive system and breast disorders) | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.